CLINICAL TRIAL: NCT03300622
Title: Evaluation of Hospitalized Patients After Thoracic Pulmonary Resection Surgery
Brief Title: Assessment in Patients After Thoracic Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Principal Investigator, Universidad de Granada
Other Study IDs: DF0070UG
Record Dates: First submitted 2017-09-20; First posted 2017-10-03 (Actual); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Thoracic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lung cancer is the leading cause of death in men and the second in women with a 5 year survival in Europe of less than 15%. One of the methods most used for its treatment is pulmonary resection. The objective of this study is to analyze the clinical profile presented to patients after pulmonary resection.

DETAILED DESCRIPTION:
One of the most widely used methods for the treatment of lung cancer is pulmonary resection. The morbidity and mortality of pulmonary resection surgery is conditioned by both the type of intervention and the patient's condition. Functional deterioration is a risk associated with hospitalization in the elderly, with a high prevalence (35-70%) and serious consequences, since in the majority it can lead to the appearance of complications not related to the reason for admission or the specific treatment. It is very important to evaluate the clinical profile of patients after pulmonary resection in order to stablish a more specific repercussion.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted for lung resection and who sign the informed consent

Exclusion Criteria:

* Patients who did not agree to sign informed consent and those who presented other types of problems to be able to adequately carry out the assessment, such as not handling the language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and / or women of legal age who are admitted for lung resection, with the approval of the physician responsible, and who sign the informed consent
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Strength in upper and lower limbs | Baseline, up to 1 month
  Changes from baseline to postintervention during hospital stay in lower and upper limbs strength. The quadriceps and the hand-grip strength is assessed using a portable dynamometer with a standard protocol allowing three attempts on each side.

SECONDARY OUTCOMES:
Exercise capacity | Baseline, up to 1 month
  Five times sit to stand test (5STS) will be used to assess exercise capacity. 5STS is a simple assessment tool that is feasible in all healthcare settings and involves asking the patient to stand up 5 times for the shortest possible time without arm support.. Saturation and heart rate will be monitored as well as levels of dyspnea and fatigue of the patient.

OTHER OUTCOMES:
Mood | Baseline, up to 1 month
  Mood in these patients will be measured by the Hospital Anxiety and Depression Scale.
Fatigue | Baseline, up to 1 month
  Fatigue will be assessed with the Fatigue Severity Scale (FSS). The FSS is a nine-item instrument designed to assess fatigue as a symptom of a variety of different chronic conditions and disorders. The scale addresses fatigue's effects on daily functioning, and its relation to motivation, physical activity, work, family, and social life, and the answers to the problem with which they are fatigued and the degree to which the problem poses a problem for them .
Changes in quality of sleep | Baseline, up to 1 month
  changes in quality of sleep from baseline to postintervention. For this purpose, the participants are going to complete the Pittsburgh Quality of Sleep Index. This is a self-rating questionnaire with seven subscores that result in a global score between 0 and 21.
Comorbidities | Baseline
  Charlson Comorbidity Index will be used to assess the comorbidities of the patients, it is a simple and valid method of estimating risk of death from comorbid disease. It contains 19 categories of comorbidity and predicts the ten-year mortality for a patient who may have a range of co-morbid conditions. Each condition is assigned with a score of 1, 2, 3 or 6 depending on the risk of dying associated with this condition.
Nutritional status | Baseline, up to 1 month
  Nutritional status was evaluated with Mini nutritional assessment (MNA) test, that is validated to provide a single, rapid assessment of nutritional status in elderly patients in outpatient clinics, hospitals, and nursing homes. The MNA test is composed of simple measurements and brief questions that can be completed in about 10 min.
Dyspnoea | PBaseline, up to 1 month
  Changes from baseline to postintervention in dyspnoea measured with Borg Scale
Dependence | Baseline, up to 1 month
  The Barthel Index determines the degree of dependence of the patient for performing the basic activities of daily living. It is a questionnaire that consists of 10 items, and at lower score, more dependency; and higher score, more independence.
Pain | Baseline, up to 1 month
  Pain will be assessed by using the Visual Analogue Scale
Cough | Baseline, up to 1 month
  The cough will be assessed with the Leicester cough questionnaire that objectively assesses chronic cough and its effect on quality of life. It is structured in three domains: physical, psychological and social.
Pain | Baseline, up to 1 month
  Pain will be assessed by using a brief pain-specific questionnaire, Brief Pain Inventory, too.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Carmen Valenza, PT, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Department of Physical Therapy, Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided